CLINICAL TRIAL: NCT02763345
Title: The Added Value of a Mobile Application of Community Case Management on Under-5 Referral, Re-consultation and Hospitalization Rates in Malawi: a Pragmatic Stepped-wedge Cluster Randomized Trial
Brief Title: The Added Value of a Mobile Application of Community Case Management on Pediatric Referral Rates in Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Imperial College London (Other); University College Cork (Other); Lund University (Other); Mzuzu University (Unknown); Luke International Norway (Unknown)
Responsible Party: Principal Investigator, Matthew Thompson, Professor, Department of Family Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 51750
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Infectious Diseases
MeSH Terms: conditions — Communicable Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paper-based CCM (Standard Care) (Active Comparator): Children are assessed and treated according to the WHO and UNICEFs paper-based Community Case Management decision aid for Malawi for a minimum of 2 and a maximum of 7-weeks. Clinical assessment is guided by the paper-based 'Sick Child Form' presented in English, and clinical data is recorded by Health Surveillance Assistants manually in the Village Clinic Register.
  Interventions: Other: Standard care
- SL eCCM App + paper CCM (Experimental): Health Surveillance Assistants use the Supporting LIFE electronic Community Case Management App (SL eCCM App) deployed on a smartphone and replicating paper-based CCM guidelines to assess and treat children in conjunction with standard care, for a minimum of 2-weeks and maximum of 7-weeks. Clinical data is recorded in both the SL eCCM App and Village Clinic Register.
  Interventions: Other: Supporting LIFE electronic Community Case Management

INTERVENTIONS:
Other: Supporting LIFE electronic Community Case Management — The SL eCCM App is smartphone application developed to run on Android operating systems 3.0 Honeycomb and above. The SL eCCM App represents an electronic format of the WHO and UNICEFs paper-based CCM clinical decision rule, currently adopted as national policy in Malawi for assessing children presenting to village clinics with acute illness.The App includes a tap-sensitive breath counter for measuring breathing rate.
  Other Names: SL eCCM App
  Arms: SL eCCM App + paper CCM
Other: Standard care
  Arms: Paper-based CCM (Standard Care)

SUMMARY:
Community Case Management (CCM) is a clinical decision aid used by frontline Health Surveillance Assistants (HSAs) in Malawi to manage uncomplicated cases of pneumonia and malaria (amongst other conditions). Children identified has having complicated illness are urgently referred to larger health facilities better equipped to clinically manage these more complex presentations. There is evidence to suggest HSAs are missing opportunities to refer seriously ill children, and parents/caregivers are failing to comply with urgent referral recommendations when given; reducing the overall effectiveness of the CCM strategy. Use of mobile technology for deploying CCM has been demonstrated in prior research as feasible to evaluate, acceptable to health workers and parents/caregivers and improving health worker fidelity to the guidelines, but it is unknown if this translates into increased referral and referral completion rates. This trial seeks to evaluate the added value of a purpose developed mobile solution for CCM, called Supporting LIFE electronic Community Case Management (SL eCCM App) on HSA referral and parent/caregiver health seeking behavior.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers aged ≥18 years with spoken fluency in Chichewa, Tonga and Tumbuka
* Children aged ≥2 months to <5 years
* Able/willing to give voluntary verbal consent

Exclusion Criteria:

* Parents/caregivers aged <18 years
* Children aged <2 months or ≥5 years
* Children who are convulsing or unconscious/unresponsive at presentation
* Parents/caregivers unable/unwilling to give voluntary verbal consent

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6995 (Actual)
Dates: Start 2016-10; Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Health worker initiated referral of children to higher-level health facilities | at the index visit (study enrollment)
Attendance/non-attendance of parent/caregivers given urgent referral recommendation at higher-level health facilities | 7-days post-enrollment

SECONDARY OUTCOMES:
Barriers and facilitators to parent/caregiver compliance with referral recommendations | <2-weeks post-enrollment
Acceptability of the SL eCCM App to HSAs and parents/caregivers | <2-weeks post-enrollment
Household-level costs associated with healthcare seeking behavior | < 2-weeks post-enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Thompson, DPhil, Principal Investigator — University of Washington

REFERENCES:
- [Derived] Chirambo GB, Thompson M, Hardy V, Ide N, Hwang PH, Dharmayat K, Mastellos N, Heavin C, O'Connor Y, Muula AS, Andersson B, Carlsson S, Tran T, Hsieh JC, Lee HY, Fitzpatrick A, Joseph Wu TS, O'Donoghue J. Effectiveness of Smartphone-Based Community Case Management on the Urgent Referral, Reconsultation, and Hospitalization of Children Aged Under 5 Years in Malawi: Cluster-Randomized, Stepped-Wedge Trial. J Med Internet Res. 2021 Oct 20;23(10):e25777. doi: 10.2196/25777. PMID 34668872
- [Derived] Hardy V, O'Connor Y, Heavin C, Mastellos N, Tran T, O'Donoghue J, Fitzpatrick AL, Ide N, Wu TJ, Chirambo GB, Muula AS, Nyirenda M, Carlsson S, Andersson B, Thompson M. The added value of a mobile application of Community Case Management on referral, re-consultation and hospitalization rates of children aged under 5 years in two districts in Northern Malawi: study protocol for a pragmatic, stepped-wedge cluster-randomized controlled trial. Trials. 2017 Oct 11;18(1):475. doi: 10.1186/s13063-017-2213-z. PMID 29020976